# CREIGHTON UNIVERSITY SCHOOL OF DENTISTRY DEPARTMENT OF PERIODONTICS

# STUDY PROTOCOL Clinical Efficacy of easy graft Classic for the treatment of Peri-implantitis

**Protocol Number: 1015456** 

Original Protocol Issue Date: May 15, 2017

Principal Investigator: Lorenzo Mordini, DDS, MS

Creighton University School of Dentistry

**Department of Periodontics** 

2500 California Plaza, Omaha, NE 68178



Sponsor: SUNSTAR Americas, Inc.

#### **CONFIDENTIALITY STATEMENT**

This document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by federal or state law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you which is indicated as privileged or confidential.

# Contents

| PROTO | OCOL SY | NOPSIS | | 4 |
|---|---|---|---|---|
| 1.0 | ВАСКО | GROUND | | 5 |
| 2.0 | SUMN | IARY AN | D STUDY RATIONALE | 11 |
| | INVESTIGATIONAL DEVICE | | | |
| | GUIDOR® easy-graft® CLASSIC | | | |
| | GUIDO | )R <sup>®</sup> Bio-r | esorbable Matrix Barrier | 16 |
| 3.0 | STUDY | DESIGN | I | 16 |
| | 3.1 | Overall | Study Design | 16 |
| | Objectives | | | |
| | 3.3 | Subject Eligibility | | 20 |
| | | - | Inclusion Criteria | |
| | | 3.3.2 | Exclusion Criteria | 21 |
| | 3.4 | Study P | Procedures | 23 |
| | | | Pre-Operative Treatment | |
| | | | Study Treatments | 24 |
| | | | Other Therapy 25 Postsurgical Care | 25 |
| | 3.5 | | Assessments | |
| | | | Summary of Clinical Assessments | |
| | | 3.5.3 | Probing Depths | 29 |
| | | | O'Leary Plaque Index | |
| | | | Laboratory Assessments | |
| | 3.6 | | le of Investigational Events | |
| | | | Screening Visit (Visit 1) | |
| | | | Post op – 1 Month (Visit 4) | |
| | | 3.6.7 | 12 Months Follow up. (Visit 7) | |
| | 3.7 | | rry of Clinical Assessments (revised by UoC to meet assessn | |
| | • • • | | | |
| | 3.7 | - | raphy | |
| | <b></b> | • | Exposure 44 | |
| | | 3.7.2 | Processing 44 | |
| | | | Handling 44 | |
| | | | Radiographic assessment | |
| | | | Derivation or calculation of variable | |
| | 3.8 | Discont | tinuation of Treatment | 46 |

 INFORMATION OF Creighton University School of Dentistry Department of Periodontics

Protocol Number: CUSD2 Revision: October 22<sup>nd</sup> 2018

Original Issue Date: January 6th 2017

| 4.0 | ADVE | ADVERSE EVENTS | |
|---|---|---|---|
| | Recor | ding and Reporting Adverse Events | 46 |
| | Recor | ding Adverse Events | 47 |
| | Gradi | ng Adverse Events | 48 |
| | Assign | ning Relationship of Adverse Events to Treatment | 48 |
| | Seriou | us Adverse Events | 49 |
| | Defini | Definition of a Serious Adverse Event | |
| | SAE re | 50 | |
| 5.0 | STATISTICAL AND ANALYTICAL PLAN | | |
| | Intent | Intent to Treat Population | |
| | Safety | Safety Population | |
| | Evalua | Evaluable Population | |
| | Missi | Missing Data | |
| | Asses | sment of Safety | 53 |
| 6.0 | REGU | LATORY AND ADMINISTRATIVE REQUIREMENTS | 53 |
| | 6.1 | IRB Requirements | 53 |
| | 6.2 | Protocol Amendments | 54 |
| | 6.3 | Informed Consent | |
| ΔΡΡΕ | NDIX I: | OUESTIONNAIRES/SURVEYS | 56 |

Protocol Number: CUSD2 Revision: October 22<sup>nd</sup> 2018

# **PROTOCOL SYNOPSIS**

| Protocol Number | 1015456 |
|---|---|
| Title | A STUDY TO DETERMINE EFFICACY OF EASY GRAFT CLASSIC FOR THE TREATMENT OF PERI-IMPLANTITIS |
| Subject Population | Subjects with history of Moderate to Severe Peri-implantitis |
| Objectives | TO ASSESS THE EFFECTVENESS OF EFFICACY OF EASY GRAFT CLASSIC |
| Number of Subjects | Maximum of 15 subjects |
| Number of Sites | Maximum 20 implants |
| Safety Endpoints | Assessments of subject safety will be based upon tabulations of the incidence of adverse events. |
| Efficacy Endpoints | Stability and health of the attachment apparatus at 6 and 12 months by measuring: Change from baseline in probing depth Change from baseline in clinical attachment level Change from baseline in width of the keratinized tissue Change from baseline in radiographic A) bone regeneration; B) pathology Esthetic satisfaction from baseline to 12 months, as assessed by both the examiner and the subject using the Visual Analog Scale (VAS), prior to and after viewing baseline photos Subject pain/discomfort questionnaire |

 $CONFIDENTIAL\ AND\ PROPRIETARY\ INFORMATION\ OF\ Creighton\ University\ School\ of\ Dentistry\ Department\ of$ 

Periodontics

Protocol Number: CUSD2 Revision: October 22<sup>nd</sup> 2018

Original Issue Date: January 6th 2017

This study will be "case series". Two periodontists will perform surgical

procedures and record surgical measurements. The blinded examiner will

perform all other clinical assessments. 15 subjects will be enrolled. Written

informed consent will be obtained from each subject prior to any study related

procedures. The study will follow subjects for safety and efficacy for 12 months

after their surgical treatment.

The day of surgery will be designated as Day 0. Subjects will have a guided bone

regeneration surgery with GUIDOR® easy-graft® CLASSIC and GUIDOR®

Bioabsorbable Membrane Matrix for the implants experiencing peri-implantitis.

The surgical side will be assessed for osseous and implant surface anomalies.

Intraoperative and postoperative measurements will be made and the flap will be

closed with sutures.

1.0 BACKGROUND

**Study Design** 

Peri-implantitis is an infectious condition of the tissues around dental implants causing loss of

supporting bone and clinical signs of inflammation such as bleeding and/or suppuration on

probing). The prevalence of this disease regards almost 10% of implants and almost 20% of

 INFORMATION OF Creighton University School of Dentistry Department of

patients<sup>1,2</sup>. Many factors influence and increase prevalence (and the risk) of peri-implantitis.

Some of those are previous history of periodontitis, smoking, diabetes as well as the type and

frequency of follow-up care. It is worth noting that the prevalence of peri-implantitis varies

depending on the parameters used in scientific papers. Bone loss and/or probing depth

threshold may vary among different authors modifying the case definition.

Different clinical protocols for treatment of peri-implantitis have been proposed, including

mechanical debridement, the use of antiseptics and local or systemic antibiotics, as well as

surgical access and regenerative procedures. Several attempts to combine the data of the

available literature in a meta-analysis have failed in the past due to insufficient data.<sup>3,4,5,6,7,8</sup>

Mombelli et all, in their review<sup>9</sup> noted that almost all studies on the treatment of peri-

implantitis in humans do not satisfy the strict criteria for a randomized controlled trial (RCT).

The main limitation was the absence of a true control group (no treatment or placebo). Trials at

the highest level of evidence compared test procedures, both of which had an unclear

<sup>1</sup> Mombelli A, Müller N, Cionca N. The epidemiology of periimplantitis. Clin Oral Implants Res 2012;23(suppl 6):67–76.

<sup>&</sup>lt;sup>2</sup> Lee CT, Huang YW, Zhu L, Weltman R. Prevalences of peri-implantitis and peri-implant mucositis: systematic review and meta-analysis. J Dent. 2017 Jul;62:1-12. doi: 10.1016/j.jdent.2017.04.011. Epub 2017 May 3. Review.

<sup>&</sup>lt;sup>3</sup> Klinge B, Gustafsson A, Berglundh T. A systematic review of the effect of anti-infective therapy in the treatment of peri-implantitis. J Clin Periodontol 2002;29(suppl 3):213–225; discussion 232–213.

<sup>&</sup>lt;sup>5</sup> Renvert S, Roos-Jansaker AM, Claffey N. Non-surgical treatment of peri-implant mucositis and peri-implantitis: A literature review. J Clin Periodontol 2008;35:305–315.

<sup>&</sup>lt;sup>6</sup> Renvert S, Polyzois I, Claffey N. Surgical therapy for the control of peri-implantitis. Clin Oral Implants Res 2012;23(suppl 6):84–94.

<sup>&</sup>lt;sup>7</sup> Muthukuru M, Zainvi A, Esplugues EO, Flemmig TF. Non-surgical therapy for the management of peri-implantitis: A systematic review. Clin Oral Implants Res 2012;23(suppl 6):77–83.

<sup>&</sup>lt;sup>8</sup> Esposito M, Grusovin MG, Worthington HV. Treatment of periimplantitis: What interventions are effective? A Cochrane systematic review. Eur J Oral Implantol 2012;5(suppl):s21–s41.

<sup>9</sup>Mombelli A, Moene R, Decaillet F. Surgical treatments of periimplantitis. Eur J Oral Implantol 2012;5(suppl):s61–s70

outcome. As it is difficult to recruit sufficient numbers of patients with peri-implantitis to take

part in a true randomized trial, some studies may have been underpowered.

In terms of outcomes, there is inconsistency about primary treatment goals and minimally

required observation periods. A recent Cochrane systematic review <sup>10</sup> included nine

randomized controlled trials in an attempt to identify the most effective interventions for

treating peri-implantitis around osseointegrated oral implants. The authors concluded that

there is no reliable evidence suggesting which could be the most effective interventions for

treating peri-implantitis. A review by Heitz-Mayfield and Mombelli<sup>11</sup> covered reports that

evaluated the effect of treatment, regardless if they were randomized trials or not. The

available evidence does not provide specific recommendations or standard protocol for peri-

implantitis treatment. Successful treatment outcomes at 12 months were reported in a

majority of patients in 7 studies. Despite favorable short-term outcomes were reported in many

studies, failure of treatment, progression or recurrence of disease and implant loss were

reported too. The main limitation of systematic reviews is the heterogeneity in study design,

length of follow-up, and exclusion/inclusion criteria.

. .

<sup>10</sup>Esposito M, Grusovin MG, Worthington HV. Interventions for replacing missing teeth: Treatment of peri-implantitis. Cochrane Database Syst Rev 2012:1

<sup>11</sup>Heitz-Mayfield and Mombelli. The therapy of peri-implantitis: a systematic review. Int J Oral Maxillofac Implants. 2014;29 Suppl:325-45. doi: 0.11607/jomi.2014 suppl

 INFORMATION OF Creighton University School of Dentistry Department of

Daugela et al<sup>12</sup> reported that in case of evident bone loss and pocket formation deeper than 5

mm, the surgical treatment seemed to be the only effective one in managing peri-implantitis

defect. Surgical regenerative treatment resulted in predictable improvement of peri-implant

clinical and radiographic parameters although this statement is limited on available studies

without proper control arm, as at the time there is a lack of controlled studies comparing

effectiveness of surgical regenerative and non-regenerative procedures to support scientific

evidence if regenerative procedures provide better outcomes.

Currently there is a lack of clear recommendation regarding choice of biomaterials for peri-

implant bone regeneration due to high heterogeneity among the studies. From the clinical

point of view, surgical regenerative treatment is a relevant treatment option of intrabony

defect component in addition to pre- and postsurgical hygiene maintenance phases and

successful implant surface decontamination. Regenerative procedures, with the application of

bone graft materials in combination or not with barrier membranes seem to give consistent

results in the term of hard and soft tissues healing of the peri-implantitis defect.

Regenerative treatment of peri-implantitis lesions can be performed in cases with considerable

pocket formation and bone loss after the acute infection has been resolved and proper oral

hygiene has been instituted. Reported clinical studies indicate that considerable bone

regeneration and re-osseointegration can be obtained by using various types of bone graft

materials and membranes. Meta-analysis of latest systematic literature review xi revealed that

<sup>12</sup>Daugela P, et alSurgical Regenerative Treatments for Peri-Implantitis: Meta-analysis of Recent Findings in a Systematic Literature Review. J

 INFORMATION OF Creighton University School of Dentistry Department of

the weighted mean of marginal bone level change was 1.97 mm, PD reduction was 2.78 mm

and BOP reduced by 52.5% by treatment with regenerative treatment. However, a different

compatibility between bone grafting material and chemically and mechanically decontaminated

implant surface might bring a different clinical outcome.

As far as the use of alloplastic grafting material, only two papers were identified in the

literature. Roos-Jansåker et al. 13, 14 evaluated regenerative treatment of peri-implantitis

comparing a bone substitute with or without a barrier membrane. Peri-implant defects were

treated with a phytogenic calcium carbonate bone substitute (Algipore) or with the bone

substitute and a resorbable synthetic membrane (Osseoquest). Successful treatment outcome

(no PD ≤ 5 and no further bone loss 12mo after treatment) was on 93% of patient treatment

with bone substitute and membrane and 89% of patients treated with bone substitute only.

Schwarz et al 15 filled peri-implant defects with either a synthetic nano-

crystalline hydroxyapatite (Ostim) or a bovine-derived xenogenic bone mineral (BioOss), and

covered with a collagen membrane (Bio-Gide). Within the limits of the present case series they

concluded that at 12 months after surgery both therapies resulted in clinically important PD

reductions and CAL gains.

Oral Maxillofac Res 2016: 9 (3): e15

<sup>13</sup>Roos-Jansåker A-M, Renvert H, Lindahl C, Renvert S. Surgical treatment of peri-implantitis using a bone substitute with or without a resorbable membrane: A prospective cohort study. J Clin Periodontol 2007;34:625–632.

<sup>14</sup>Roos-Jansåker A-M, Lindahl C, Persson GR, Renvert S. Long-term stability of surgical bone regenerative procedures of peri-implantitis lesions in a prospective case-control study over 3 years. J Clin Periodontol 2011;38:590–597.

<sup>15</sup> Healing of intrabony peri-implantitis defects following application of a nanocrystalline hydroxyapatite (Ostim) or a bovine-derived xenograft (Bio-Oss) in combination with a collagen membrane (Bio-Gide). A case series. Schwarz F, Bieling K, Latz T, Nuesry E, Becker J J Clin Periodontol. 2006 Jul;33(7):491-9.

 INFORMATION OF Creighton University School of Dentistry Department of

Due to scarcity of literature on the use of alloplast on peri-implant treatment, the purpose of

the study is to assess the effectiveness of the novel in-situ hardening β -TCP material, Easy-

Graft® CLASSIC and polylactide based biodegradable membrane, GUIDOR® Biodegradable

Matrix Barrier, following clinically adequate decontamination procedures. The author thinks

that the specific properties of this grafting material may favor treatment of peri-implantitis. A

recent study by Canullo<sup>16</sup> et al. analyzed the efficacy of Easy-Graft® CLASSIC on the treatment of

peri-implantitis. After removal of granulomatous tissue and decontamination of the titanium

exposed implant surface, Easy-Graft was placed on the defect as a protection from soft tissue

invasion. The authors noted a pronounced increase in mucosal recession and clinical

attachment level with stable peri-implant conditions at six and 12 months. Plaque index,

bleeding on probing and probing depths values were significantly reduced at six and 12 months.

Radiographic analysis demonstrated from partial to complete filling of the defect in all of the

cases at six and 12 months.

Easy-graft remains moldable until it comes in contact with blood or tissue fluids. When the

material is soaked in blood in bone defects it hardens in a few minutes to form stable porous

scaffold for bone regeneration. This characteristic of graft material gives better handling for the

clinician. The hardening of the material could provide an increased stability of the blood clot

around implant defect and favor hard tissue deposition and maturation. The Easy-Graft®

CLASSIC manufacturer recommends GUIDOR® Bioabsorbable Membrane Matrix to be used

<sup>16</sup> Canullo L, Peñarrocha Oltra D, Tallarico M, Aloy Prosper A, Chocer H, Peñarrocha Diago M. Surgical treatment of circumferential and semicircumferential defects due to periimplantitis: a prospective case series cohort study. J Oral Science Rehabilitation.

2016 Dec;2(4).

 INFORMATION OF Creighton University School of Dentistry Department of

simultaneously in order to maximize its effects. The main difference between this proposed

study and Canullo's will be the use of GUIDOR® Bioabsorbable Membrane Matrix in conjunction

with Easy-Graft® CLASSIC

The authors of this present study considered the outcome of the peri-implant surgical therapy

successful if: implant survival with no peri-implant probing depths (PD) ≥ 5 mm, with

concomitant bleeding on probing (BOP) and no suppuration, in addition to no additional or

progressive bone loss. If these criteria were met, it can be assumed that no further intervention

other than nonsurgical maintenance care would be required, and the treatment outcome

would therefore be regarded as successful.

2.0 **SUMMARY AND STUDY RATIONALE** 

The present study was designed to demonstrate the EFFICACY OF EASY GRAFT CLASSIC FOR

THE TREATMENT OF PERI-IMPLANTITIS.

 INFORMATION OF Creighton University School of Dentistry Department of

Periodontics


Easy-graft® CLASSIC, is commercially available alloplastic bone graft granules consists of

pure  $\beta$  -TCP, which has been commonly used for the indication of ridge preservation <sup>17, 18</sup>,

peri-implant bone augmentation<sup>19</sup>, sinus elevation<sup>20</sup> and other treatment of intraoral /

maxillofacial osseous defects<sup>21</sup>. It has unique handling capacity based on an extremely thin

coating of the graft granules with poly(lactic-co-glycolic acid) (PLGA). PLGA is used as a raw

material to manufacture dental membranes, suture materials and resorbable screws.

Before application, the granules are mixed with BioLinker® which consists of water and N-

Methyl-2-pyrrolidone (NMP). It is non-volatile solvent which has been in used in various

medical products for more than 10 years. Easy-graft remains moldable until it comes in

contact with blood or tissue fluids. When the material is soaked in blood in bone defects it

hardens in a few minutes to form stable porous scaffold for bone regeneration. This

characteristic of graft material gives better handling for the clinician.

Regenerative treatment of peri-implantitis lesions can be performed in cases with

considerable pocket formation and bone loss after the acute infection has been resolved

and proper oral hygiene has been instituted. Reported clinical studies indicate that

 $^{17}$  Leventis MD, et.al. (2016) Minimally invasive alveolar ridge preservation utilizing an in situ hardening  $\beta$ -tricalcium phosphate bone substitute. A multicenter case series. Int J Dent. ID 5406736

10 of the state of

<sup>18</sup> Schneider D, et.al. (2014) Labial soft tissue volume evaluation of different techniques for ridge preservation after tooth extraction: a randomized controlled clinical trial. J Clin Periodontol. 41(6): 612-617.

<sup>19</sup> El Sayed et. al. (2015) After socket preservation of upper anterior teeth. Alexandria Dental Journal. 40: 79-85

<sup>20</sup> Troedhan A, et.al. (2015) Biomechanical Stability of Dental Implants in Augmented Maxillary Sites: Results of a Randomized Clinical Study with Four Different Biomaterials and PRF and a Biological View on Guided Bone Regeneration. BioMed Res Int. ID

850340

<sup>21</sup> Neumeyer S. et al. (2010) The use of polylactide-coated ß-TCP: Closure of oro-antral communications. Implants. 4:32-36

 INFORMATION OF Creighton University School of Dentistry Department of

considerable bone regeneration and re-osseointegration can be obtained by using various

types of bone graft materials and membranes. Meta-analysis of latest systematic literature

review<sup>22</sup> revealed that the weighted mean of marginal bone level change was 1.97 mm, PD

reduction was 2.78 mm and BOP reduced by 52.5% by treatment with regenerative

treatment. However, a different compatibility between bone grafting material and

chemically and mechanically decontaminated implant surface might bring a different clinical

outcome. The purpose of the study is to assess the effectiveness of in-situ hardening  $\beta$  -

TCP material, easy-graft CLASSIC, for the regenerative treatment of peri-implantitis with

polylactide based biodegradable membrane (GUIDOR® Bio-resorbable Matrix Membrane)

following clinically adequate decontamination procedures.

The day of surgery will be designated as Day 0. Subjects will have periodontal surgery based

on the protocol of Guided Bone Regeneration. Subjects will have a guided bone

regeneration surgery with GUIDOR® Bio-resorbable Matrix Membrane and Easy graft classic

for the implants experiencing peri-implantitis. The surgical side will be assessed for osseous

and implant surface anomalies. Intraoperative and postoperative measurements will be

made and the flap will be closed with sutures.

<sup>22</sup> Daugela P, et al. (2016) Surgical regenerative treatment for peril-implantitis: Meta-analysis of recent findings in a systematic

literature review. J Oral Maxillofac Res. 9 (3): e15

 INFORMATION OF Creighton University School of Dentistry Department of

The preliminary phase of the study will comprise completion of medical and dental

histories, signing of consent forms, obtaining radiographs and photographs, performing

screening assessments to confirm eligibility, and instruction in oral hygiene techniques.

Before the periodontal surgical procedure, subjects may undergo plaque removal, then root

planing and scaling to the areas to be treated, if such treatment is indicated. The final

esthetic outcome of the treated sites will be evaluated by the patients using the Visual

Analog Scale (VAS) ranging from "Very Unsatisfied" to "Very Satisfied" (before and after

viewing baseline photos). Other clinical assessments will include: subject pain/discomfort

questionnaire, change in probing depth, change in clinical attachment level, change in width

of keratinized tissue from baseline to 6 and 12 months and change in radiographic bone

gain and pathology. Digital photographs will be obtained at each study visit and

radiographs of the test sites will be made at the baseline, 6 and 12 month visits.

The primary efficacy parameters will include:

Esthetic satisfaction from baseline to six months of all treated areas, as assessed by

both the examiner and the subject using the Visual Analog Scale (VAS), prior to and

after viewing baseline photos

Subject pain/discomfort questionnaire

Change from baseline in probing depth (PD) measured from the mucosal margin to

the bottom of the probeable pocket

Gingival recession (Rec) measured from the implant platform (IP) to the mucosal

margin

Change from baseline visit in clinical attachment level (CAL) measured from IP to the

bottom of the probeable pocket

Change from baseline in width of the keratinized tissue (KT)

• Change from baseline in radiographic a) bone gain; b) pathology

**INVESTIGATIONAL DEVICE** 

GUIDOR® easy-graft® CLASSIC

GUIDOR® easy-graft® CLASSIC is bone grafting system contains: syringe containing beta-

tricalcium phosphate (β-TCP) granules coated with poly (lactide-co-glycolide) (PLGA) and

ampule containing BioLinker® Activator (N-methyl-2-pyrrolidone and water).

Easy-graft CLASSIC is a bio-resorbable, synthetic, porous bone graft substitute. It consists of

two components: granules (supplied in syringe) and BioLinker activator (supplied in ampule).

After mixing the components together, easy-graft CLASSIC forms a moldable mass that can be

applied directly from the syringe into the bone defect. Easy-graft CLASSIC hardens in contact

with body fluids, allowing a working time of approximately one minute after application into

the bone defect. Easy-graft CLASSIC is provided in the particle size of  $500 - 1000 \mu m$ . The

scaffold is a biocompatible and osteoconductive that allows for complete resorption by the

 INFORMATION OF Creighton University School of Dentistry Department of

body. β-TCP and PLGA are derived from synthetic raw materials. Easy-graft CLASSIC comes

sterilized via gamma irradiation.

**GUIDOR®** Bio-resorbable Matrix Barrier

GUIDOR® Matrix Barrier are made of polylactic acid with a citric acid ester. It is double-

layered; the external layer has large rectangular perforations which face the overlying soft

tissues and permit connective tissue infiltration, while the inner layer has small circular

perforations which face bone and inhibit fibrous tissue ingrowth. It maintains its barrier

function for 6 weeks at least, with complete resorption occurring by 6 months. Available

membrane dimensions are 15 mm x 20 mm or 20 mm x 28 mm. The membrane is provided in

a transparent plastic tray in a sealed aluminum pouch. It comes sterilized via e-beam.

3.0 STUDY DESIGN

3.1 Overall Study Design

This study will be case series, with two periodontists and an examiner. Both of the

periodontists will perform surgical procedures and record surgical measurements. The

blinded examiner will perform all other clinical assessments. 15 subjects will be enrolled.

Written informed consent will be obtained from each subject prior to any study related

procedures.

 INFORMATION OF Creighton University School of Dentistry Department of

The study will follow subjects for safety and efficacy for 6 and 12 months after their surgical

treatment.

Screening will take place no more than 32 days prior to the first treatment and will include

the clinical assessments required to confirm eligibility. Clinical photograph, radiographs of

the implant treated, clinical measurements will be taken and recorded (Pocked Depth,

Mucosal Recession, Clinical Attachment Level). Two to four (2-4) weeks prior to the first

study treatment, subjects may undergo plaque removal and root planing and scaling to the

areas to be treated, if appropriate. Also, they will receive personalized oral hygiene

instructions to reach full-mouth plaque score (FMPS) <20% and full-mouth bleeding score

(FMBS) <20%, which will be considered requirement for surgery to occur.

The day of surgery will be designated as Day 0. Subjects will have peri-implant regeneration

surgery.

If possible, implant crown will be removed with attention not to damage it. Healing screw

will be placed on the implants. Upon flap elevation and debridement of the peri implant

lesion, the operator will record the type of bony defect associated to the treated implant

(see Inclusion criteria 3). Titanium Implant surface will be debrided with rotating burs and

brushes (PERI-SET Swden&Martina Inc.), and decontaminated with EDTA

(Straumann PrefGel. pH neutral, 24% EDTA) for 2 minutes and with the alternation of

Perio-Flow Chlorhexidine mouthwash (GUM® ParoEx®, Chlorhexidine Gluconate Oral Rinse

USP 0,12%, SUNSTAR) saline water and  $H_2O_2$  using cotton pellets. After the completion of

these procedures, Easy-graft® CLASSIC will be placed to fill the peri-implant defect.

 INFORMATION OF Creighton University School of Dentistry Department of

GUIDOR® Bio-resorbable Matrix Membrane will be placed on top of the easy-graft classic. If

the implant crown was successfully removed and healing screw placed, the implant will be

covered by the flap and submerged. Intraoperative and postoperative measurements will

be made and the flap will be closed with sutures. Patients will be instructed to take 500 mg

of amoxicillin three times a day for 7 days, starting at least one hour prior the procedure.

Fifteen (15) male or female subjects, aged 21 to 85 years, will be recruited for the study

from existing patient databases, as well as, from screenings of volunteers responding to

advertisements, if necessary.

**Objectives** 

The objectives of this study are to assess the EFFICACY OF EASY GRAFT CLASSIC FOR THE

TREATMENT OF PERI-IMPLANTITIS.

3.2.1 Primary Efficacy Endpoints

Change from baseline in probing depth

Change from baseline in clinical attachment level

Change from baseline in width of the keratinized tissue

Change from baseline in radiographic a) bone gain; b) pathology

Esthetic satisfaction from baseline to six months of all treated areas, as assessed by

both the examiner and the subject using the Visual Analog Scale (VAS), prior to and

after viewing baseline photos

 INFORMATION OF Creighton University School of Dentistry Department of

Subject pain/discomfort questionnaire

## 3.2.2 Study Duration

The duration of this study is to be twelve (12) months following the surgical procedure.

# 3.2.3 Study Timeline Summary

| | Deceline | Post | Post | Post | Post | Post |
|---|---|---|---|---|---|---|
| Screening | Baseline<br>and Surgery | Treatment | Treatment | Treatment | Treatment | Treatment |
| | | Evaluation | Evaluation | Evaluation | Evaluation | Evaluation |
| Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 |
| Within 32 | | | | | | |
| days | Day 0 | Week 1 | Month 1 | Month 3 | Month 6 | Month 12 |
| of surgery | | ± 3 days | ±7 days | ± 14 days | ± 14 days | ± 14 days |

# 3.2.4 Safety Endpoints

Assessments of subject safety will include a tabulation of the incidence of adverse events. All treatment-related adverse events that occur up to 30 days excepting surgery related AEs within 48 hours after any treatment will be recorded, and all serious adverse events throughout the study will be recorded.

 INFORMATION OF Creighton University School of Dentistry Department of

Periodontics

Protocol Number: CUSD2 Revision: October 22<sup>nd</sup> 2018 3.3 Subject Eligibility

3.3.1 Inclusion Criteria

Subjects must meet the following inclusion criteria to be eligible for the study:

1. Subject has read and signed the IRB approved consent form before treatment.

2. Subject must be age 21 or above.

3. Subject must be willing and able to follow study procedures and instructions.

4. Subject affected by moderate to severe peri-implant disease\*.

5. Treated chronic periodontitis and proper periodontal maintenance care,

Dental implant must meet the following criteria to be selected for the study:

1. Implant presenting PD ≥ 6 mm

2. Radiographic implant bone loss more than 25% of the implant length (Apex of the implant

to implant platform)<sup>23</sup>.

3. Peri implant bone defect being a buccal dehiscence and semicircular bone resorption to the

middle of the implant body, buccal dehiscence and circular bone resorption with lingual

bone plate intact or circular bone resorption with buccal and lingual bone plates intact

<sup>23</sup> Froum SJ, Rosen PS. A proposed classification for peri-implantitis. Int J Periodontics Restorative Dent. 2012 Oct;32(5):533-40.

 INFORMATION OF Creighton University School of Dentistry Department of

4. Single tooth implant restoration or implant supported fixed partial denture.

3.3.2 Exclusion Criteria

Subject with any of the following will not be eligible for the study:

Subjects participating (currently or within 30 days prior to enrollment) in other clinical

trials involving therapeutic intervention (either medical or dental).

• Subjects with poor oral hygiene as indicated by a score of greater than 50% on the

O'Leary Plaque Index.

• Subjects with a systemic condition, which would preclude periodontal treatment,

including but not limited to uncontrolled diabetes.

• Subjects with acute infectious lesions in the areas intended for treatment.

Subjects taking chronic (i.e., > 2 weeks), therapeutic doses of medications known to

affect bone metabolism such as nonsteroidal anti-inflammatory drugs or

bisphosphonates. Prophylactic aspirin (≤ 325 mg q.d.) for cardiovascular indications will

be permitted in subjects.

Female subjects who are pregnant or lactating, or sexually-active female subjects who

are of childbearing potential and are not using hormonal or barrier methods of birth

control. (except for when a result of pregnancy test is negative)

• Subjects who are on any chronic antibiotic or steroidal therapy.

 INFORMATION OF Creighton University School of Dentistry Department of

• Smoker using more than 10 cigarettes or equivalent per day.

• Smoker using cigar, smokeless tobacco use or e-cigarette.

• Subjects diagnosed with drug induced gingival hyperplasia (e.g. calcium channel

blockers).

• Subjects with radiographic evidence of pathology in other areas of the mouth besides

implant area to be treated.

• Implant mobility.

• Subjects with parafunctional habits and not wearing bite guard.

•

3.3.3 Investigator Training and Qualification

The investigator(s) will be trained before participation in the study during a site initiation by

means of a detailed description of all study procedures including the methods of obtaining

study endpoints (measurements). The examiner will be calibrated so that the difference is 1

mm or less between his or her measurements and the principal investigator. Each examiner

will measure the recession depth on two subjects three times each during each calibration

session. These measurements will be recorded on a case report form and analyzed to

ensure each examiner's accuracy is 1 mm or less. Examiner recalibration will be performed

at the six month follow-up visit to ensure that his or her accuracy in measuring recession

depth remains within that limit. Any examiner who has greater than 1.0 mm variability

 INFORMATION OF Creighton University School of Dentistry Department of

from the principal investigator will undergo retraining by the principal investigator, as

necessary.

One examiner will make all the measurements for each subject. The investigator

guarantees that the examiner, who has working experience with the probe, is well qualified.

All investigators will be noted on the Investigator's Agreement and appropriate

qualifications (CV and license) will be maintained in the investigator file.

3.3.4 Blinding and Probe Calibration

All study staff, with the exception of the treating clinician will be blinded to the treatment

administered. Only calibrated UNC 15 probes will be used.

3.4 Study Procedures

3.4.1 Pre-Operative Treatment

Medical examination and past history as well as dental examination and past history will

be completed at this stage.

Within 32 days prior to surgery, the subject will undergo plaque removal and the test sites

will be undergo to root planing and scaling (if determined to be appropriate treatment by

the investigator). Two to four (2-4) weeks prior to the first study treatment, subjects may

undergo plaque removal and root planing and scaling to the areas to be treated, if

 INFORMATION OF Creighton University School of Dentistry Department of

Periodontics


appropriate. Also, they will receive personalized oral hygiene instructions to reach full-

mouth plaque score (FMPS) <20% and full-mouth bleeding score (FMBS) <20%, which will

be considered requirement for surgery to occur.

3.4.2 Study Treatments

Screening will take place no more than 32 days prior to the first treatment and will include

the clinical assessments required to confirm eligibility. Informed Consent Form will be

signed at Screening Visit (Visit 1). Clinical photograph, radiographs of the implant treated,

clinical measurements will be taken and recorded (Pocked Depth, Mucosal Recession,

Clinical Attachment Level).

The day of surgery will be designated as Day 0. Subjects will have peri-implant regeneration

surgery.

Whenever possible implant crown will be removed and cleaned. Healing screw will be

placed on the implant. Upon flap elevation and debridement of the peri implant lesion, the

operator will record the type of bony defect associated to the treated implant (see Inclusion

criteria 3). Titanium Implant surface will be debrided with rotating burs and brushes (PERI-

SET, Sweden&Martina Inc.), and decontaminated with EDTA (PrefGel: Straumann) for 2

minutes and with the alternation of Perio-Flow Chlorhexidine mouthwash (GUM® ParoEx®,

Chlorhexidine Gluconate Oral Rinse USP 0,12% SUNSTAR), saline water and H2O2 using

cotton pellets. After the completion of these procedures, Easy-graft® CLASSIC will be placed

on the peri-implant defect surface. GUIDOR® Bio-resorbable Matrix Membrane will be

 INFORMATION OF Creighton University School of Dentistry Department of

placed on top of the easy-graft classic and stabilized. If the implant crown was successfully

removed, flaps will be primary closed and the implant will be covered completely. Second

stage, minimally invasive surgery to gain access to the implant will be performed at 6

months. Intraoperative and postoperative measurements will be made and the flap will be

closed with sutures. Patients will be instructed to take 500 mg of amoxicillin three times a

day for 7 days, starting at least one hour prior the procedure.

Fifteen (15) male or female subjects, aged 21 to 85 years, will be recruited for the study

from existing patient databases, as well as, from screenings of volunteers responding to

advertisements, if necessary.

3.4.3 Other Therapy

No other dental therapies are permitted in conjunction with the study treatments, dental

emergencies excluded (i.e. Acute abscesses, Pulpitis, tumors or oral lesions).

3.4.4 Postsurgical Care

Patients will be instructed to take 500 mg of amoxicillin three times a day for 7 days,

starting at least one hour prior the procedure. In case of allergy to amoxicillin, patient will

assume 300mg Clindamycin three times a day for 7 days. Subjects will be advised to follow

good oral hygiene habits in all non-study sites by brushing twice daily using a soft bristled

toothbrush, and flossing once per day. All subjects will be instructed to avoid brushing and

avoid the use of interdental cleaning devices for the first seven days following the surgical

 INFORMATION OF Creighton University School of Dentistry Department of

procedure. In addition, all subjects will be instructed to avoid chewing directly on the test

sites and to avoid trauma to the test sites for the first week following the surgery. During

that interval, the subjects will be instructed to rinse twice daily after meals with 0.12%

chlorhexidine gluconate non-alcohol oral rinse. After the first week, the subjects will be

instructed to resume gentle tooth brushing and interdental cleaning with dental floss and

continue the 0.12% chlorohexidine gluconate oral rinse for the first 4 weeks following

surgery. All subjects will receive local implant cleaning at the month 3, 6 and 12 follow up

visits.

3.4.5 Management of Post-Surgical Oral Pain

Any pre-surgical pain medications should be recorded and noted as such (i.e. pre-surgical

pain medication). Post-surgical pain can be divided into mild, moderate, and severe levels

and requires a subjective assessment by the periodontists based on knowledge of the

surgical procedure performed and the presenting signs and symptoms of the subject. Pain

as a secondary outcome to an adverse event, such as infection, is to be excluded if pain is an

expected outcome of such events. Treatment of the pain is usually the best indicator of

pain intensity.

MILD (Over-the Counter)

Acetaminophen 250 or 500 mg.

Products include: Tylenol<sup>®</sup>, Datril<sup>®</sup>, Anacin<sup>®</sup>3

Ibuprofen

 INFORMATION OF Creighton University School of Dentistry Department of

Products include: Motrin® 800 mg

MODERATE (Prescription Only)

Tylenol<sup>®</sup> No. 3 (codeine and acetaminophen)

Vicodin® (hydrocodone 5 mg and acetaminophen 500 mg)

Vicodin ES<sup>®</sup> (hydrocodone 7.5 mg and acetaminophen 750 mg)

Lortab® (hydrocodone 5 mg, 7.5 mg, 10 mg and acetaminophen 500 mg)

SEVERE (Prescription Only)

Demerol® 50 mg (Meperidine)\*

Percocet® or Tylox® (oxycodone 5 mg and acetaminophen 500 mg)\*

\*Triplicate prescription where applicable

3.4.6 Post-surgical Control, Professional Tooth Cleaning, Maintenance Care.

The objective of the post-operative appointments for professional tooth cleaning is both the

removal of plaque and staining from the treated areas and the monitoring of the healing

events. Post-surgical controls and professional tooth cleaning will be performed at s 3, 6

and 12 months post-surgical. At these appointments, the conditions of the soft tissue at the

treated sites will be evaluated. The overall level of oral hygiene will be evaluated and

reinstruction will be given as needed at all visits.

Instructions on post-operative care will be repeated at each appointment. In particular, the

following points should be covered during the first month: (1) continue chlorhexidine rinses

 INFORMATION OF Creighton University School of Dentistry Department of

(from surgery to four weeks post-op); (2) resume gentle brushing; and (3) avoid vigorous

chewing on, or trauma to, the treated areas.

At week 6, subjects will be instructed to gradually resume interproximal cleaning, as well as

chewing, in the treated areas. All subjects will be maintained by full mouth professional

prophylaxis and calculus removal once every three months, excluding surgical sites which

will be maintained supragingivally.

All treatment-related adverse events that occur up to 30 days excepting surgery related AEs

within 48 hours after any treatment will be recorded in CRFs, and all serious adverse events

throughout the study will be recorded.

3.5 Clinical Assessments

3.5.1 Summary of Clinical Assessments

All examinations and measurements will be performed in accordance with the Schedule of Events.

Data will be collected and assessments will be made on study sites treated.

3.5.2 Primary Efficacy Assessment

• Esthetic satisfaction from baseline to 6 and 12 months of all treated areas, as assessed by both

the examiner and the subject using the Visual Analog Scale (VAS), prior to and after viewing

baseline photos

Subject pain/discomfort questionnaire

 INFORMATION OF Creighton University School of Dentistry Department of

Change from baseline in probing depth

Change from baseline visit in clinical attachment level

Change from baseline visit in width of the keratinized tissue

Change from baseline in radiographic a) bone gain; B) pathology

3.5.3 Probing Depths

Clinical probing depths of the periodontal sulcus will be measured using the a UNC 15 periodontal

probe. Measurements will be performed without local anesthesia at six (6) locations around each

study tooth. The number of additional locations to be measured around each experimental site will

be determined by the extent and morphology of the area. Interproximal pocket depths will be

recorded at the deepest point probable at the contact points from both buccal and lingual aspects.

Buccal and lingual pocket depth measurements will be recorded at the mid-buccal and mid-lingual

sites. All pocket depth measurements will be rounded down to the nearest mm and recorded. In

conjunction with recording the pocket depths, any bleeding from the periodontal pockets will be

indicated by marking an asterisk on the figure recorded for the depth measurement for that same

pocket.

3.5.4 O'Leary Plaque Index

The plaque index is determined by scoring the percentage of individual tooth surfaces with plaque.

The following procedure will be followed:

Apply disclosing solution to all exposed tooth surfaces.

 INFORMATION OF Creighton University School of Dentistry Department of

Rinse to remove any excess solution.

Examine each tooth surface (mesial, distal, facial, lingual) at the dento-gingival junction for presence of plaque.

Presence of plaque at the dento-gingival junction is indicated by making a dash in the appropriate spaces on the plaque control record diagram (see Figure 1).

If a tooth is missing, draw a line through the tooth on the diagram. Missing teeth should not be counted in the total number of surfaces scored.

Calculate the plaque index by dividing the number of surfaces with plaque by the total number of surfaces scored, and then multiply by 100 to obtain a percentage.

Figure 1 Plaque Control Record

#### 3.5.5 Laboratory Assessments



The following laboratory assessments will be conducted at screening:

Urine pregnancy test (females of child-bearing potential only)

 INFORMATION OF Creighton University School of Dentistry Department of Periodontics

Protocol Number: CUSD2 Revision: October 22<sup>nd</sup> 2018

Original Issue Date: January 6<sup>th</sup> 2017

#### 3.6 Schedule of Investigational Events

## 3.6.1 Screening Visit (Visit 1)

At the screening visit the following procedures and assessments will be performed within 32 days prior to surgery:

- Informed Consent
- Subject registration
- Medical history collection and physical examination:
  - Record of past therapy
  - Urine pregnancy test (females of child-bearing potential only)
  - Medications
- Dental history collection
  - Record of past therapy
- Screening assessments to determine eligibility:
  - O'Leary Plaque Index
  - Probing depths
  - Implant mobility,
  - Clinical attachment level
  - Obtain baseline radiographs of study sites

#### Dental cleaning

 INFORMATION OF Creighton University School of Dentistry Department of

Oral hygiene instruction

• Supragingival plaque control, as appropriate

• Examiner and subject baseline esthetic satisfaction VAS assessments

Radiographs of all target study sites

3.6.2 Baseline/Treatment (Visit 2)

Visit 2 may occur concurrently with Visit 1. If separate visits are to occur, Visit 2 must occur within

32 days of the screening examine.

• Examiner calibration (for first 2 subjects enrolled only)

Preoperative and Intraoperative digital photographs

Concomitant medications

Surgical procedure

Post-operative instructions

• Collection of any Adverse Events

3.6.3 Post op - Week 1 (Visit 3)

An Investigator will rate and record the judgment of healing

• Study personnel will obtain clinical photographs of surgical sites taking care not to place apical

tension on flap

 INFORMATION OF Creighton University School of Dentistry Department of

• Post-operative instructions (e.g. Chlorhexidine rinse) and pain management according to

standard procedures

Complete Pain Rating Scale

Rate and record color and texture of treated areas

Adverse event review

Concomitant medication review

Suture removal according to healing

Measurement of width of keratinized tissue

Pain Medication review

3.6.4 Post op – 1 Month (Visit 4)

Rate and record the color and texture of treated areas

Digital photographs

Rate and record judgment of healing

Clinical attachment level

• The examiner and subject esthetic satisfaction VAS assessments (before and after viewing

baseline photos)

Supragingival plaque control as indicated

Oral hygiene instruction

Complete pain rating scale

Concomitant medications

 INFORMATION OF Creighton University School of Dentistry Department of

Collection of Adverse Events

• Pain medication review

3.6.5 3-Months Follow up (Visit 5)

At the month 3 visit (Day 90 ± 14 days) the following procedures and assessments will be

performed:

Rate and record the color and texture of treated areas

Digital photographs

Rate and record judgment of healing

Measurement of width of keratinized tissue

Clinical attachment level

• The examiner and subject esthetic satisfaction VAS assessments (before and after viewing

baseline photos)

Supragingival plaque control as indicated

Oral hygiene instruction

• Complete pain rating scale

Concomitant medications

Collection of Adverse Events

Pain medication review

Implant area professional cleaning

3.6.6 6 Months Follow up. (Visit 6)

Subjects will return to the clinic for a study visit 6 months (± 14 days) after surgery. The following

procedures and assessments will be performed at this visit:

Digital photographs

Radiographs of all treated sites

The examiner and subject esthetic satisfaction VAS assessments (before and after viewing

baseline photos)

Rate and record the color and texture of treated areas

Rate and record judgment of healing

Measurement of width of keratinized tissue

Clinical attachment level

Supragingival plaque control as indicated

Oral hygiene instruction

Complete pain rating scale

Concomitant medications

Probing depth

Collection of Adverse Events

Pain medication review

Adverse Events review

Implant area professional cleaning

3.6.7 12 Months Follow up. (Visit 7)

Subjects will return to the clinic for a study visit 6 months (± 14 days) after surgery. The following

procedures and assessments will be performed at this visit:

Digital photographs

Radiographs of all treated sites

The examiner and subject esthetic satisfaction VAS assessments (before and after viewing

baseline photos)

Rate and record the color and texture of treated areas

Rate and record judgment of healing

Measurement of width of keratinized tissue

Clinical attachment level

Supragingival plaque control as indicated

Oral hygiene instruction

Complete pain rating scale

Concomitant medications

Probing depth

Collection of Adverse Events

Pain medication review

Adverse Events review

Implant area professional cleaning
 INFORMATION OF Creighton University School of Dentistry Department of Periodontics
Protocol Number: CUSD2
Revision: October 22<sup>nd</sup> 2018

Original Issue Date: January 6<sup>th</sup> 2017 

3.7 Summary of Clinical Assessments (revised by UoC to meet assessment for implant tooth)

All examinations and measurements will be accomplished in accordance with the Schedule of

Procedures (See Study Flowchart).

Oral Hygiene Status

Plaque recorded as present (1) or not present (0) on buccal and lingual surfaces of study teeth only

Bleeding following Angulated Probing

Bleeding will be registered at the surgical sites by means of pulling a probe with 60° angle to the

root surface along the gingival margin.

**Probing Pocket Depth** 

Distance of probe penetration (UNC 15 periodontal probe), measured from the gingival margin to

the bottom of the probable pocket of the buccal surface to the nearest 0.5 mm.

**Probing Proximal Pocket Depth** 

 INFORMATION OF Creighton University School of Dentistry Department of

Periodontics

Distance of probe penetration (UNC 15 periodontal probe), measured from the gingival margin to

the bottom of the probable pocket of the mesial and distal surface to the nearest 0.5 mm.

Clinical Attachment Level (CAL)

Distance of probe penetration (UNC 15 periodontal probe) measured from fixed reference point to

the nearest 0.5 mm.

**Proximal Probing Attachment Loss** 

Distance of probe penetration (UNC 15 periodontal probe) measured from fixed reference point at

the mesial and distal aspect of the tooth to the nearest 0.5 mm.

**Recession Depth** 

The distance between the fixed reference point and the soft tissue margin, measured to the

nearest 0.5 mm with a UNC 15 periodontal probe. At the 6 and 12 month visit, tissue coronal to

the fixed reference point will be recorded as a negative measurement

 INFORMATION OF Creighton University School of Dentistry Department of

Periodontics

Width of Keratinized Tissue

The distance between the free gingival margin and the muco-gingival junction, measured to the

nearest 0.5 mm with a graded periodontal probe. To facilitate the identification of the muco-

gingival line, a probe may be used horizontally to move the mucosa in a coronal direction, creating

a fold at the muco-gingival junction. Shiller's Iodine Solution may also be used to identify the

muco-gingival junction

**Examination of Defects During Surgery** 

After the flaps have been raised and the area debrided, characterization of the morphology and

measurements of the defects are made, with the UNC 15 periodontal probe, and recorded as

follows:

Alveolar Bone Level (Before and after osteoplasty if needed)

Notation of intra marrow penetration of alveolar crest

Notation of alveolar crest topography and whether osteoplasty was to be performed to refine

contours.

 INFORMATION OF Creighton University School of Dentistry Department of

Periodontics

**Clinical Photographs** 

Clinical photographs will be taken of each tooth involved in the study before, during and after

surgery, at Weeks 1, and 6 post surgery and at the 3, and 6 month follow-up examinations.

Post-Op Discomfort and Satisfaction Questionnaires

The subject's satisfaction with respect to postoperative discomfort between test and

control quadrants will be evaluated by asking the subject about pain, bleeding,

swelling and sensitivity using 10 cm visual analogue scale (See Appendix 1).

| | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 |
|---|---|---|---|---|---|---|---|
| | Screen | | | | | | |
| | 0-32 Days | | Post-op | 1 Month | Month 3 | Month 6 | Month 12 |
| Procedure/ Assessment | Prior | Day 0 | Day 7 | 42± 7 Days | 90± 14 Days | ±14 Days | ±14 Days |
| | Surgery | | | | | | |
| Informed Consent | Х | | | | | | |
| Eligibility/ Study Lesion Identification, | X | | | | | | |
| Subject Registration | ^ | | | | | | |
| Demographics/Dental/Medical History | X | | | | | | |
| O'Leary Plaque Index | X | | | | | X | X |
| Probing Depths | X | | | | | X | X |
| Pregnancy Test | X <sup>1</sup> | | | | | | |
| Radiographic Exam | X | | | | | X | X |
| Dental Cleaning | X | | | | X | X | x |

| Digital Photos | | X | Х | X | X | X | X |
|---|---|---|---|---|---|---|---|
| Examiner and Subject GORS and VAS of | | x | x | X | X | x | X |
| esthetic satisfaction | | ^ | ^ | ^ | ^ | <b>A</b> | <b>A</b> |
| Plaque Control/Oral Hygiene Instruction | X | х | X | X | X | X | X |
| Concomitant Medications | X | х | X | X | X | X | X |
| Adverse Events | | Х | Х | X | X | X | X |
| Clinical Attachment level | X | | | | | X | X |
| Examiner calibration | | Х | | | | | |
| Easy Graft Classic surgery | | х | | | | | |
| Second stage surgery for submerged | | | | | | x | |
| implants only | | | | | | ^ | |
| Rate and record Judgment of Healing | | | X | x | X | X | X |
| Pain Rating Scale | | | X | X | x | X | X |
| Color and Texture | | | X | X | X | X | X |
| Width of Keratinized Tissue | | | | X | X | X | X |
| 1. In | females | <u> </u> | of | child-b | earing | potent | ial |

 INFORMATION OF Creighton University School of Dentistry Department of Periodontics

Protocol Number: CUSD2

Original Issue Date: January 6th 2017

only

3.7 Radiography

Radiographs will be taken using a modified Rinn system in order to obtain radiographs with

minimum projection error. Rinn system is a radiograph sensor holder that favors a standard

system to have reproducible radiograph images. We will customize this holder in order to

reproduce standard radiographic image. Evaluable bitewings radiographs will be taken in

each of the tooth regions included in the study.

3.7.1 Exposure

Intraoral film, 24 × 40 mm, from the same batch will be used.

3.7.2 Processing

Digital X-ray system will be used.

3.7.3 Handling

Study radiographs are stored in Axium system.

3.7.4 Radiographic assessment

Intra-oral biewing radiographs will be obtained at baseline, at 6 and 12 months. These

radiographs should be taken using device to standardize during course of the study and

should image the target tooth and at least 2 mm on either side of the osseous defect.

 INFORMATION OF Creighton University School of Dentistry Department

of Periodontics

Protocol Number: CUSD2

Original Issue Date: January 6th 2017


The following standardizing technique will produce repeatable diagnostic quality

radiographs with close to identical geometry and image clarity.

Once the exposure parameters are selected they should not be changed during the

course of the study. Send the image files to the central reading center at each study site

for analysis following the instructions.

3.7.5 Derivation or calculation of variable

Image processing software is used to capture measurements (MiPACS Dental

Enterprise). Measurement tool will be calibrated with a 1 millimeter radiographic image.

The measurements are taken from a stationary landmark (Distal and Mesial portion of

implant platform - Bdp and Bmp) to the mesial and distal bone crest of osseous defect in

millimeters (Bda and Bma). In order to calculate percentage of bone fill (or residual

defect) this last measured will be compared with implant length noted on the chart.

Subsequent images are logged in and saved to the file. Linear measurements of bone

height along root surfaces are made using the same method as the original defect.

• Linear bone change (distal) =  $Bd_{p(0.6.12)} - Bd_{a(0.6.12)}$ 

Linear bone change (mesial) =  $Bm_{p(0,6,12)} - Bm_{a(0,6,12)}$ 

Where (0.6.12) is the measure at baseline, 6 and 12 months.

 INFORMATION OF Creighton University School of Dentistry Department

of Periodontics

3.8 Discontinuation of Treatment

Subjects may be withdrawn from the study prior to completion of treatment for the

following reasons:

Subject withdrawal of consent

Investigator's decision

Death

Poor maintenance of oral hygiene

Lack of compliance

Discontinues Orthodontics treatment and/or other treatments on study site(s) and

adjacent teeth

When a subject is terminated from the study prior to completion of treatment, the

subject will continue to be evaluated as scheduled. Attempts will be made to

perform all follow-up assessments and procedures required by the protocol.

4.0 ADVERSE EVENTS

**Recording and Reporting Adverse Events** 

An Adverse Event (AE) is defined as any untoward medical occurrence in a subject of a

clinical investigation administered an investigational product and that does not necessarily

have a causal relationship with this treatment. An AE can therefore be any unfavorable and

unintended sign (including an abnormal laboratory finding), symptom, or disease temporally

 INFORMATION OF Creighton University School of Dentistry Department

of Periodontics

Protocol Number: CUSD2

associated with the use of an investigational product, whether or not related to use of the

product.

**Recording Adverse Events** 

All adverse events occurring after surgical procedure will be collected during the entire trial.

Each adverse event will be followed until the adverse event has resolved or stabilized.

During visits, subjects should be encouraged to report adverse events spontaneously or in

response to general, non-directed questioning.

Standard medical terminology for the AE and the associated body system

Description of adverse event and clinical consequences

Date and time of onset

Date and time of resolution of the adverse event

Whether or not the event is ongoing

Severity of the event

Relationship between the adverse event and the investigational agent or related

procedure

Description of any therapy administered and associated outcome (actions required)

Outcome of the AE

Whether or not the effect was serious and/or unanticipated

All AEs, regardless of seriousness, severity, or presumed relationship to study

therapy, must be recorded using medical terminology in the source document and

on the adverse event case report form.

 INFORMATION OF Creighton University School of Dentistry Department

of Periodontics

Protocol Number: CUSD2

Original Issue Date: January 6th 2017

Whenever possible, a diagnosis should be given when signs and symptoms are due

to common etiology (e.g., cough, runny nose, sneezing, sore throat, and head

congestion should be reported as "upper respiratory infection").

Each adverse event should be reported separately. For example, "nausea and

vomiting" should be recorded as two (2) separate events.

**Grading Adverse Events** 

Common Terminology Criteria for Adverse Events v3.0, (on the NCI website,

http://ctep.info.nih.gov) will be used to grade all toxicities/adverse events. Adverse events

not included in the CTCAE v.3.0 should be reported with common medical terminology and

graded according to definitions in the CTC Manual.

Assigning Relationship of Adverse Events to Treatment

A relationship must be assigned by the investigator to each reported adverse event, and will

be documented as follows:

• Unrelated The event is clearly due to causes other than the study treatment.

• Unlikely Toxicity is doubtfully related to the study treatment. The event was

most likely related to other factors such as the subject's clinical state,

concomitant drugs or other therapeutic interventions.

• Possible The event follows a reasonable temporal sequence from the time of

study treatment administration, but could have been produced by

 INFORMATION OF Creighton University School of Dentistry Department

of Periodontics

Protocol Number: CUSD2

other

factors such as the subject's clinical state, therapeutic interventions

or

concomitant drugs.

Probable

The event follows a reasonable temporal sequence from the time of

study treatment, and follows a known response pattern to treatment.

The toxicity cannot be reasonably explained by other factors such as

the subject's clinical state, therapeutic interventions or concomitant

drugs.

• Definite

The event follows a reasonable temporal sequence from the time of

study treatment administration, follows a known response pattern to

the study treatment, cannot be reasonably explained by other factors

such as the subject's condition, concomitant drugs or therapeutic

interventions, AND either occurs immediately following

administration of the study treatment, improves on stopping the

study treatment, or reappears on re-exposure.

**Serious Adverse Events** 

**Definition of a Serious Adverse Event** 

A Serious Adverse Event (SAE) is defined as any event meeting any of the following criteria:

 INFORMATION OF Creighton University School of Dentistry Department

of Periodontics

Protocol Number: CUSD2

Original Issue Date: January 6th 2017

Is life-threatening or fatal

Requires, or significantly prolongs, inpatient hospitalization

Results in persistent or significant disability and/or incapacity

Is a congenital anomaly or birth defect

Requires medical or surgical intervention to prevent one of the outcomes listed

above

**SAE** report to Sponsor and IRB

Investigators and other study site personnel must inform appropriate Sponsor

representatives of any SAE that occurs during the course of the study within one day

(i.e., immediately but no later than the end of the next business day) of when he or she

becomes aware of it.

The Sponsor representative will work with the Investigator to compile all the necessary

information and ensure that the appropriate Sponsor personnel receives a report by day

one for all fatal and life-threatening cases and by day five for all other SAEs.

If an AE becomes a SAE, this and other relevant follow-up information must also be

provided to Sponsor within one day for all fatal and life-threatening cases and by day

five for all other SAEs.

 INFORMATION OF Creighton University School of Dentistry Department

of Periodontics

Protocol Number: CUSD2

The Investigator is responsible for informing the ethics committee of SAEs as per local

requirements.

SUNSTAR IS RESPONSIBLE FOR INFORMING THE REGULATORY AUTHORITY OF DEVICE RELATED SAES AS PER

REQUIREMENTS.

5.0 STATISTICAL AND ANALYTICAL PLAN

Intent to Treat Population

The primary efficacy analysis and summaries will be performed on the "intent to treat" (ITT)

population, defined as all subjects who successfully completed the screening to enter this

trial.

**Safety Population** 

All safety summaries and analyses will be performed on the safety population, defined to be

all subjects.

**Evaluable Population** 

All secondary efficacy analyses will be performed on an evaluable population, defined to be

all subjects who received surgical treatment in accordance with the protocol.

 INFORMATION OF Creighton University School of Dentistry Department

of Periodontics

Protocol Number: CUSD2

Original Issue Date: January 6th 2017


Subjects exiting after undergoing surgery, but before month 6 due to treatment-related

adverse events will be included in the evaluable population. Subjects that do not complete

the assessments due to satisfaction with treatment will also be included in the evaluable

population. All attempts will be made to collect complete follow-up evaluations for these

subjects despite study exit. These subjects will be included in the analysis based on the

assessments that are completed.

Subjects will be deemed non-evaluable if they do not meet the eligibility criteria as outlined

in the protocol. Other reasons to be considered non-evaluable include protocol violations,

as described below, and any actions that compromise the effectiveness of the treatment,

for non-efficacy or safety related reasons.

Protocol violators consist of subjects who do not comply with the protocol in terms of

treatment administration, visit timing, and/or assessment compliance. Each protocol

violation will be discussed between Investigators and the Sponsor to evaluate the impact on

the statistical assessment before performing the analyses.

**Missing Data** 

It is not anticipated that many subjects will exit the study prematurely or will miss visits. The

reasons for early termination, along with the timing of the early terminations will be

provided.

Subjects missing a baseline evaluation will be discussed between Investigators and the

Sponsor to evaluate the impact on the statistical assessment before performing the

analyses

 INFORMATION OF Creighton University School of Dentistry Department

of Periodontics

Protocol Number: CUSD2

**Assessment of Safety** 

Adverse events with an onset within 30 days of any surgical treatment will be recorded and

tabulated. All adverse events will be tabulated by first occurrence of the event, maximum

severity, and strongest relationship to study treatment by body system.

6.0 REGULATORY AND ADMINISTRATIVE REQUIREMENTS

6.1 **IRB Requirements** 

United States Federal regulations require that all investigational studies be conducted

under the auspices of an Institutional Review Board (IRB), as defined in the Code of Federal

Regulations, Title 21, Part 56. This committee, the makeup of which must conform to the

Federal, State and local guidelines regarding such, will approve all aspects of the Study,

including said Protocol and Informed Consents to be used, prior to initiation. The formal

written approval notice must be signed by the chairman or authorized designee and must

identify the specific protocol. In cases where an IRB member has a conflicting interest,

abstention of that individual from voting should be documented. The investigator will

provide the sponsor with a copy of the communication from the Committee to investigator

indicating approval of the protocol and consent form. All changes to the protocol and

consent form must be reviewed and approved prior to implementation, except where

necessary to eliminate apparent immediate hazards to human subjects.

 INFORMATION OF Creighton University School of Dentistry Department

The investigator must also report to the IRB, at least annually, on the progress of the

investigation. Continuing IRB review should be documented by a letter from the IRB.

Notification to the IRB by the investigator within three months after completion,

termination, or discontinuation of the study at the specific site must be documented.

6.2 **Protocol Amendments** 

Amendments will originate from the sponsor and will be provided to the investigator for

submission to his or her IRB for its review and approval prior to implementation. It should

be noted that when an amendment to a protocol substantially alters the study design or

increases potential risk to the study subject, the informed consent should be revised and if

applicable, subject's consent to continue participation should again be obtained.

No deviations from the protocol should be made except in emergency situations where

alternative treatment is necessary for the protection, proper care and wellbeing of subjects.

In situations requiring a departure from the protocol, the investigator or other physician in

attendance will contact the sponsor's clinical representative by fax or telephone. If

possible, this contact will be made before implementing any departure from the protocol.

In all cases, contact with the sponsor's clinical representative must be made as soon as

possible in order to discuss the situation and agree on an appropriate course of action. The

case report form and source document will describe any departure from the protocol and

the circumstances requiring it.

 INFORMATION OF Creighton University School of Dentistry Department

of Periodontics

6.3 Informed Consent

In accordance with the Code of Federal Regulations, Title 21, Part 50.20 the investigator will

be responsible for obtaining an Informed Consent, signed by the subject or legally

authorized representative, from every subject prior to his/her participation in the study.

The consent form that is used must be the current version and must be approved by both

the reviewing IRB and by the sponsor. Informed consent will be obtained from the subject

after a full explanation of the purpose of the study, risks and discomforts involved, potential

benefits, etc. have been provided by the investigator both verbally and in writing. The

original signed copy of the informed consent must be maintained in the institution's

records, and is subject to inspection by a sponsor representative.

## APPENDIX I: QUESTIONNAIRES/SURVEYS

- 1. Examiner's Judgment of Healing
- 2. Pain Visual Analogue Scales
- 3. Discomfort and Satisfaction Questionnaire
- 4. Color and Texture Scale
- 5. Inflammation Score

 INFORMATION OF Creighton University School of Dentistry Department of Periodontics

Protocol Number: CUSD2

Original Issue Date: January 6th 2017 

#### **EXAMINER'S JUDGMENT OF HEALING**

| 1 | circl | Δ | rac | $n \cap $ | nca |
|---|-------|---|-----|--------------|------|
| ١ | | | 103 | $\mathbf{p}$ | 1136 |

| Uppe | r Righ | nt Qua | adrant: |
|------|--------|--------|---------|
|------|--------|--------|---------|

| Much worse | Worse than | | Better than | Much better |
|---------------|------------|-------------|-------------|---------------|
| than expected | expected | As Expected | expected | than expected |

# Upper Left Quadrant:

| Much worse | Worse than | | Better than | Much better |
|---------------|------------|-------------|-------------|---------------|
| than expected | expected | As Expected | expected | than expected |

Lower Right Quadrant:

 INFORMATION OF Creighton University School of Dentistry Department

of Periodontics

Protocol Number: CUSD2

Original Issue Date: January 6th 2017


| Much worse | Worse than | | Better than | Much better |
|---------------|------------|-------------|-------------|---------------|
| than expected | expected | As Expected | expected | than expected |

Lower Left Quadrant:

| Much worse | Worse than | | Better than | Much better |
|---------------|------------|-------------|-------------|---------------|
| than expected | expected | As Expected | expected | than expected |

of Periodontics

Protocol Number: CUSD2

Original Issue Date: January 6th 2017 

#### **PAIN VISUAL ANALOGUE SCALES**

| Please have po | atient complete the scales below by drawing a single vertical lin | e across each scale at |
|---|---|---|
| the point corre | esponding to the patient's level of pain. | |
| | Upper Right Quadrant | |
| No Pain | | Extreme Pain |
| | Upper Left Quadrant | |
| No Pain | | Extreme Pain |
| | Lower Right Quadrants | |
| No Pain | | Extreme Pain |

 INFORMATION OF Creighton University School of Dentistry Department

of Periodontics

Protocol Number: CUSD2

Original Issue Date: January 6th 2017 

## Lower Left Quadrant

| | <del></del> |
|---------|--------------|
| No Pain | Extreme Pain |

## **DISCOMFORT & ESTHETIC SATISFACTION QUESTIONNAIRE: Maxillae**

| Category | Right Quadrant | Left Quadrant |
|-------------|----------------|---------------|
| Sensitivity | None | None |
| | Mild | Mild |
| | Moderate* | Moderate* |
| | Severe* | Severe* |
| | Duration: | Duration: |
| Bleeding | None | None |
| | Mild | Mild |
| | Moderate* | Moderate* |
| | Severe* | Severe* |

 INFORMATION OF Creighton University School of Dentistry Department of Periodontics

Protocol Number: CUSD2

Original Issue Date: January 6th 2017 

| | | 1 |
|---|---|---|
| | Duration: | Duration: |
| Swelling | None | None |
| | Mild | Mild |
| | Moderate* | Moderate* |
| | Severe* | Severe* |
| | Duration: | Duration: |
| (*Record as Adverse Event) | | |
| Has the patient experience | ed any other differences betwee | en the Left and Right Study sites? |
| □ Y □ N | | |
| If Yes, explain: | | |
| Overall, how satisfied is t | ne patient with the <b>appearance</b> | of the study sites? |
| Right Study Site | | |
| □ Very Satisfied □ Satis | fied Neither Unsatisfied | □ Very Unsatisfied |
| Left Study Site | | |
| □ Very Satisfied □ Satis | fied Neither Unsatisfied | □ Very Unsatisfied |
| If not satisfied, please exp | olain: | |
| | e patient experience the most di | |
| Examiner's signature: | | Date: |

 INFORMATION OF Creighton University School of Dentistry Department

of Periodontics

Protocol Number: CUSD2

Original Issue Date: January 6th 2017  Color and texture will be scored in relation to adjacent tissues as follows:

#### **DISCOMFORT & SATISFACTION QUESTIONNAIRE: Mandible**

| Category | Right Quadrant | Left Quadrant |
|-------------|----------------|---------------|
| Sensitivity | None | None |
| | Mild | Mild |
| | Moderate* | Moderate* |
| | Severe* | Severe* |
| | Duration: | Duration: |
| Bleeding | None | None |
| | Mild | Mild |
| | Moderate* | Moderate* |
| | Severe* | Severe* |
| | Duration: | Duration: |
| Swelling | None | None |
| | Mild | Mild |
| | Moderate* | Moderate* |
| | Severe* | Severe* |
| | Duration: | Duration: |

## (\*Record as Adverse Event)

 INFORMATION OF Creighton University School of Dentistry Department of Periodontics

Protocol Number: CUSD2

Original Issue Date: January 6th 2017

| Has the patient experienced any other differences between the Left and Right Study sites? |
|---|
| □ Y □ N |
| f Yes, explain: |
| Overall, how satisfied is the patient with the appearance of the study sites? |
| Right Study Site |
| □ Very Satisfied □ Satisfied □ Neither □ Unsatisfied □ Very Unsatisfied |
| Left Study Site |
| □ Very Satisfied □ Satisfied □ Neither □ Unsatisfied □ Very Unsatisfied |
| f not satisfied, please explain: |
| Overall, which side did the patient experience the most discomfort? Right Left |
| Examiner's signature:Date: |

 INFORMATION OF Creighton University School of Dentistry Department of Periodontics

Protocol Number: CUSD2

Original Issue Date: January 6th 2017 